CLINICAL TRIAL: NCT02904902
Title: A Phase 3 Multicenter, Open-label, Single Arm Study of the Safety and Efficacy of Adalimumab in Japanese Subjects With Moderate to Severe Hidradenitis Suppurativa
Brief Title: Open-label Study of Adalimumab in Japanese Subjects With Hidradenitis Suppurativa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-573
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Hidradenitis Suppurativa
Keywords: efficacy; safety; adalimumab; japanese participants
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adalimumab (Experimental): Open-label adalimumab 160 mg subcutaneous injection at Week 0 (Baseline), 80 mg at Week 2, and 40 mg every week starting at Week 4. After Week 52, Participants who consent to receive the 80 mg eow dose, will switch from 40 mg ew to 80 mg eow at Week 0x (80 mg eow period until the end of the study).
  Interventions: Drug: adalimumab

INTERVENTIONS:
Drug: adalimumab — Subcutaneous Injection
  Other Names: Humira

SUMMARY:
This study investigates efficacy, safety and pharmacokinetics of adalimumab in Japanese subjects with moderate to severe hidradenitis suppurativa (HS).

DETAILED DESCRIPTION:
Prior to initiation of this study, global Phase 2b study and pivotal Phase III studies were completed in the Western countries and market authorization of adalimumab was approved in United States (US) and European Union (EU) for the treatment of subjects with HS. The differences between this study and global studies include sample size, study design, duration, and race.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a diagnosis of HS;
* Participant must have any HS symptom at least 6 months prior to Baseline;
* HS lesions must be present in at least 2 distinct anatomic areas, one of which must be Hurley Stage II or Hurley Stage III;
* Participant must have stable HS for at least 2 months (60 days) prior to Screening and also at the Baseline visit;
* Participant must have a total abscess and inflammatory nodule (AN) count of greater than or equal to 3 at the Baseline visit.

Exclusion Criteria:

* Prior treatment with adalimumab or other anti-tumor necrosis factor (TNF) therapy or participation in adalimumab trial;
* Any other active skin lesion or condition that may interfere with assessment of HS;
* Participants received antibiotic treatment for HS within 28 days prior to the Baseline visit other than those allowed per protocol. Participant on permitted oral antibiotic treatment (doxycycline or minocycline only) for HS who have not been on a stable dose for at least 28 days prior to the Baseline visit;
* Participants received prescription topical therapies for the treatment for HS within 14 days prior to the Baseline visit;
* Participants received systemic non-biologic therapies with potential therapeutic impact for HS less than 28 days prior to the Baseline visit;
* Participants received oral concomitant analgesics (non-opioids and opioids) for HS-related pain within 14 days prior to the Baseline visit.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (8):
- Japan (8):
  - Nagoya City University Hospital /ID# 151495, Nagoya, Aichi-ken
  - Kurume University Hospital /ID# 152579, Kurume-shi, Fukuoka
  - Takagi Dermatological Clinic /ID# 151906, Obihiro, Hokkaido
  - University of the Ryukyus Hosp /ID# 152268, Nakagami-gun, Okinawa
  - NHO Osaka National Hosp /ID# 152452, Osaka, Osaka
  - Tokai University Hachioji Hosp /ID# 151338, Hachiōji, Tokyo
  - Tokyo Medical University Hospital /ID# 154171, Shinjuku-ku, Tokyo
  - Fukuoka University Hospital /ID# 151350, Fukuoka

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/adalimumab_M15-573.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab: Open-label adalimumab 160 mg subcutaneous injection at Week 0 (Baseline), 80 mg at Week 2, and 40 mg every week starting at Week 4.
Period: Overall Study
Arm/Group | Adalimumab
Started | 15
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (6.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Modified Sartorius Scale [Mean (Standard Deviation); unit: units on a scale] — The Sartorius Scale is used to quantify the severity of HS. Points are awarded for 12 body areas. The total Sartorius Scale is the sum of the 12 regional scores. Scale scores range from 0 to infinite, with larger scores representing higher severity of HS. Baseline is defined as the last non-missing value on or before the date of the first dose of study drug.
  units on a scale | 137.3 (59.21)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Hidradenitis Suppurativa Clinical Response (HiSCR) at Week 12
Description: HiSCR is defined as at least a 50% reduction in the total abscess and inflammatory nodule (AN) count with no increase in abscess count and no increase in draining fistula count relative to Baseline.
Time Frame: Week 12
Population: Full Analysis Set: all participants from sites that complied with Good Clinical Practice and received at least 1 dose of study drug and had at least 1 post-treatment efficacy assessment. Non responder imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 15
percentage of participants | 86.7 [59.5 to 98.3]

2. Secondary Outcome: Percentage of Participants Achieving AN Count of 0, 1, or 2 at Week 12
Description: The percentage of participants with AN counts lowered to 0, 1, or 2 at Week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 15
percentage of participants | 73.3 [44.9 to 92.2]

3. Secondary Outcome: Percentage of Participants Achieving at Least 30% Reduction and at Least 1 Unit Reduction From Baseline in Patient's Global Assessment of Skin Pain (NRS30) - At Worst at Week 2 Among Participants With Baseline Numeric Rating Scale (NRS) >=3
Description: The participant's Global Assessment of Skin Pain NRS was used to assess the worst skin pain due to HS. Scores range from 0 (no skin pain) to 10 (skin pain as bad as you can imagine). The assessments were completed on a daily diary by participants before they went to bed and responded to the items based on a recall period of the "last 24 hours."
Time Frame: Week 0 (Baseline), Week 2
Population: Full Analysis Set: all participants from sites that complied with Good Clinical Practice and received at least 1 dose of study drug and had at least 1 post-treatment efficacy assessment. Participants with Baseline NRS - at worst >=3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 9
percentage of participants | 33.3 [7.5 to 70.1]

4. Secondary Outcome: Change From Baseline to Week 12 in Modified Sartorius Scale Score
Description: The Sartorius Scale is used to quantify the severity of HS. Points are awarded for 12 body areas (left and right axillae, left and right sub/inframammary areas, intermammary area, left and right buttocks, left and right inguino-crural folds, perianal area, perineal area, and other). For each area, points are awarded for nodules (2 points for each); abscesses (4 points); fistulas (4 points); scars (1 point); longest distance between two lesions (2-6 points, 0 if no lesions); and if lesions are separated buy normal skin (yes-0 point; no-6 points). The total Sartorius Scale score is the sum of the 12 regional scores. Scale scores range from 0 to infinite, with larger scores representing higher severity of HS.
Time Frame: Baseline (last non-missing value on or before the date of first dose of study drug), Week 2, Week 4, Week 8, Week 12
Population: Full Analysis Set: all participants from sites that complied with Good Clinical Practice and received at least 1 dose of study drug and had at least 1 post-treatment efficacy assessment. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 15
units on a scale
  Week 2 | -16.7 (15.06)
  Week 4 | -38.7 (31.46)
  Week 8 | -49.9 (48.10)
  Week 12 | -61.4 (45.05)

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 70 days after the last dose of study drug. The mean duration of adalimumab exposure was 717.5 days (median 742.0 days, range 112 - 883 days).
Arm/Group | Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 5/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (N=15)
Cellulitis (Infections and infestations) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (N=15)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Dermoid cyst (Congenital, familial and genetic disorders) | 1 (1)
Asthenopia (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Dental caries (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Gastric polyps (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2)
Injection site induration (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Swelling (General disorders) | 2 (2)
Xerosis (General disorders) | 1 (1)
Erythrasma (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 6 (6)
Nasopharyngitis (Infections and infestations) | 5 (10)
Paronychia (Infections and infestations) | 1 (1)
Periodontitis (Infections and infestations) | 4 (4)
Postoperative wound infection (Infections and infestations) | 1 (1)
Pulpitis dental (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Tinea infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Lymphocyte count increased (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (4)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (2)
Nail pigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
Wisdom teeth removal (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT02904902/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT02904902/SAP_001.pdf